# Statistical analysis of cross-sectional survey

# 1. Descriptive Statistics:

- **Demographics:** Frequencies and percentages for categorical variables (e.g., surgeon specialty, years of experience) and measures of central tendency (mean, median) and dispersion (standard deviation, interquartile range) for continuous variables.
- Survey Responses: Frequencies, percentages, and summary statistics for responses to closed-ended questions.

## 2. Reliability Analysis:

- **Internal Consistency:** Cronbach's alpha will be calculated to assess the reliability of multi-item scales.
- Test-Retest Reliability: If applicable, test-retest reliability will be evaluated using intraclass correlation coefficients (ICCs).

#### 3. Inferential Statistics:

- Comparative Analysis:
  - Chi-Square Tests: To compare categorical variables between different groups (e.g., comparing responses between surgeons from low vs.high volume centers).
  - t-Tests/ANOVA: To compare means of continuous variables between two or more groups

## Regression Analysis:

- Linear Regression: To predict continuous outcomes based on independent variables
- Logistic Regression: To predict binary outcomes based on independent variables.

# 4. Multivariate Analysis:

- **Factor Analysis:** To identify underlying factors from the survey items related to planning and technical aspects.
- **Cluster Analysis:** To identify distinct groups of surgeons based on their responses.

# 5. Qualitative Analysis:

- Thematic Analysis: For open-ended responses, thematic analysis will be conducted to identify common themes and patterns.
- **Content Analysis:** To quantify the presence of certain themes or keywords in open-ended responses.

### 6. Handling Missing Data:

- **Imputation Methods:** Multiple imputation or other appropriate methods will be used to handle missing data.
- **Sensitivity Analysis:** To assess the impact of missing data on the results.

## 7. Statistical Software

• The analysis will be conducted using SPSS and R.

## 8. Ethical Considerations

• **Informed Consent:** Participants will provide informed consent before participating in the survey.

# Statistical analysis of PMSG planning study

#### 1. Descriptive Statistics:

 Means, standard deviations, and ranges for the coordinates of the central points of the fenestrations (angle degrees and

- distance from the proximal margin of stent fabric) and for the diameters of the 4 fenestrations will be calculated.
- Summary statistics for the percentage of surface overlap between corresponding fenestrations will be provided.

# 2. Paired t-tests or Wilcoxon Signed-Rank Tests:

 Depending on the normality of the data (which will be be checked using Shapiro-Wilk test), paired t-tests (for normally distributed data) or Wilcoxon signed-rank tests (for non-normally distributed data) to compare the central points' coordinates and diameters of the fenestrations between the study PMSG plannings and control PMSG.

# 3. Regression Analysis:

• Linear regression analysis to examine the relationship between the participant-designed and template-designed measurements, identifying any systematic bias.

## 4. Graphical Methods:

- Scatter plots to visually compare the coordinates and diameters of the fenestrations between the two methods.
- Box plots to visualize the distribution of differences in the measurements.

#### 5. Statistical Software

The analysis will be conducted using SPSS and R.

# Statistical analysis of Delphi Rounds

#### 1. Data Collection

• **Instrument:** Structured questionnaires with rating Likert scale ranging from 1 to 5, where 1 indicates strong disagreement and 5 indicates strong agreement.

#### 2. Data Coding:

Ratings are numerically coded for analysis.

## 3. Statistical Analysis

- 1. Descriptive Statistics:
  - Summary Statistics: Mean, median, standard deviation, interquartile range, and frequency distribution of ratings for each item in each round.
  - Visualization: Box plots and histograms to visualize the distribution of ratings.

### 2. Consensus Measurement:

- Interquartile Range (IQR): IQR for each item to assess the degree of consensus.
- Median Ratings: Median ratings across rounds to observe convergence towards consensus.

## 3. Stability of Ratings:

 Stability Index: Percentage of unchanged ratings between rounds for each item to measure stability and convergence.

## 4. Agreement Analysis:

Kendall's W (Coefficient of Concordance): To measure the overall agreement among panelists for each round. Values range from 0 (no agreement) to 1 (complete agreement).

- Intraclass Correlation Coefficient (ICC): To assess the reliability of ratings and the degree of agreement among panelists.
- 5. Comparison of Rounds:
  - Wilcoxon Signed-Rank Test: To compare ratings between consecutive rounds and identify significant changes.
  - Friedman Test: If there are more than two rounds, to detect differences in ratings across multiple rounds.
- 6. Handling Disagreement:
  - Analysis of Disagreement: Analysis of reasons for discordance based on qualitative feedback from panelists.
- 7. Sensitivity Analysis:
  - Outlier Analysis: Sensitivity analysis by excluding extreme ratings from outliers.

## 5. Statistical Software

• **Software Packages:** The analysis will be conducted using SPSS, R, and Stata.

## 6. Confidentiality Considerations

• **Confidentiality:** Ratings and open responses from panelists will be kept confidential to avoid risk of individual's influence and groupthink.